CLINICAL TRIAL: NCT03014674
Title: An Open Label, Randomised, Three Arm, Single Dose, Multicentre, Parallel Group Study in Healthy Subjects to Compare the Pharmacokinetics of Subcutaneous Mepolizumab When Delivered as a Liquid Drug Product in a Safety Syringe or an Auto Injector With a Reconstituted Lyophilised Drug Product From a Vial
Brief Title: A Study to Compare the Pharmacokinetics of Mepolizumab as a Liquid Drug in a Safety Syringe or an Autoinjector Versus Lyophilised Drug
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204958; 2016-002405-19 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2016-12-15; First posted 2017-01-09 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Asthma
Keywords: SB-240563; subcutaneous; lyophilized drug product; Mepolizumab; liquid drug product; safety syringe; auto injector
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Liquid mepolizumab in safety syringe (Experimental): Subjects will receive a single dose of 100 mg liquid mepolizumab administered subcutaneously using a prefilled syringe within a safety syringe according to randomization.
  Interventions: Biological: Liquid mepolizumab; Device: Prefilled Safety Syringe
- Liquid mepolizumab in an autoinjector (Experimental): Subjects will receive a single dose of 100 mg liquid mepolizumab administered subcutaneously using a prefilled autoinjector, according to randomization.
  Interventions: Biological: Liquid mepolizumab; Device: Prefilled autoinjector
- Lyophilised mepolizumab from vial (Active Comparator): Subjects will receive a single dose of 100 mg reconstituted lyophilized mepolizumab manually administered subcutaneously according to randomization
  Interventions: Biological: Lyophilized mepolizumab

INTERVENTIONS:
Biological: Lyophilized mepolizumab — Mepolizumab will be provided as white, uniform, lyophilized cake in vials with unit dose strength of 100 mg/vial for reconstitution in 1.2 mL sterile water for injection (SWFI). Following reconstitution it forms a clear to opalescent, colorless to pale yellow solution for SC injection.
  Arms: Lyophilised mepolizumab from vial
Biological: Liquid mepolizumab — Mepolizumab will be provided as a clear to opalescent, colorless to pale yellow sterile solution for SC injection, supplied in a single-use, prefilled autoinjector or safety syringe containing 100 mg/mL mepolizumab with sodium phosphate, citric acid, sucrose ethylenediaminetetraacetic acid and polysorbate 80.
  Arms: Liquid mepolizumab in an autoinjector; Liquid mepolizumab in safety syringe
Device: Prefilled autoinjector — Single use, disposable autoinjector will be assembled with the prefilled syringe containing the drug product. It will enable automatic delivery of the drug product under the power of a spring mechanism following activation of the device. Start and end of injection clicks will inform the user of correct use. A plastic needle will cover shield the needle before and after injection to minimize the potential for needle stick injuries.
  Arms: Liquid mepolizumab in an autoinjector
Device: Prefilled Safety Syringe — Single use, disposable safety syringe with a retracting needle guard and locking system.
  Arms: Liquid mepolizumab in safety syringe

SUMMARY:
Mepolizumab (SB-240563) is a humanized monoclonal antibody (Immunoglobulin G1, kappa, mAb) that blocks human interleukin-5 (hIL-5) from binding to the interleukin (IL)-5 receptor complex expressed on the eosinophil cell surface and thus inhibits signaling. This study will compare the pharmacokinetics and safety of mepolizumab administered as a liquid drug product in two different devices with the reconstituted lyophilized drug product in healthy subjects. Subjects will receive a single administration of 100 milligram (mg) mepolizumab as a single injection. The randomization will be stratified by body weight (<70 kilogram (kg), 70 <80 kg and >=80 kg) and the site of injection will be randomized 1:1:1 to the upper arm, abdomen or thigh. Approximately 243 healthy subjects will be randomized so that at least 9 subjects are randomized to each mepolizumab treatment within each weight strata and 3 subjects within each mepolizumab treatment, weight strata and injection site. Each subject will participate in the study for up to approximately 16 weeks (up to 85 days after drug administration), and will have a screening visit, a single dose treatment period, and a follow-up visit.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age and over at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or ability to interpret study results.
* Body weight >=50 kg and body mass index (BMI) within the range 19.0-30 kg/square meter(m^2) (inclusive)
* Male or Female: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: pre-menopausal females with documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up; confirmation of bilateral tubal occlusion; hysterectomy; documented bilateral oophorectomy; post- menopausal females. Subject is of reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until 16 weeks after the administration of the single dose of study medication.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol. The subject must be able to understand and communicate in the native language of the site, e.g. German in German sites.

Exclusion Criteria

* Alanine transaminase >1.5x upper limit of normal (ULN)
* Bilirubin >1.5xULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTc corrected by Fridericia's (QTcF) formula>450 milliseconds (msec)
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or 12-lead electrocardiogram.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) before the first dose of study medication and until study completion, unless in the opinion of the investigator and GlaxoSmithKline Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units for females and >21 units for males. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary nicotine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening. Limit of >500 nanogram/mL.
* Involved in any activities likely to result in any significant decrease or increase in body weight during the study period (e.g. 'crash' dieting, bodybuilding).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive test for human immunodeficiency virus antibody.
* Subjects with known, pre-existing helminthes infestation within 6 months prior to Day 1.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* A positive pre-study drug/alcohol screen.
* A vulnerable subject. Defined as individuals whose willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.
* Subjects who work for the Sponsor, contract research organization, or one of the study centers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Baltimore, Maryland, United States
- GSK Investigational Site, Berlin, Germany
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20060

REFERENCES:
- [Background] Shabbir S, Pouliquen IJ, Bentley JH, Bradford ES, C Kaisermann M, Albayaty M. The Pharmacokinetics and Relative Bioavailability of Mepolizumab 100 mg Liquid Formulation Administered Subcutaneously to Healthy Participants: A Randomized Trial. Clin Pharmacol Drug Dev. 2020 Apr;9(3):375-385. doi: 10.1002/cpdd.726. Epub 2019 Jul 17. PMID 31317668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, multi-center, open-label, parallel-group, single-dose study in healthy participants. The participants were administered one of 3 different mepolizumab treatments (a liquid drug product in a safety syringe; a liquid drug product in an autoinjector; a reconstituted lyophilized drug product from a vial).
Pre-assignment Details: A total of 246 participants were randomized and 244 participants received study treatment. Two participants were randomized in error
Groups:
- Lyophilized Vial: Participants were administered 100 milligram per milliliter (mg/mL) subcutaneous (SC) dose of mepolizumab as lyophilized powder reconstituted with sterile water for injection from vial. Participants were administered a single SC dose in upper arm, abdomen or thigh.
- Liquid Autoinjector: Participants were administered 100 mg/mL SC dose of mepolizumab liquid formulation via disposable pre-filled autoinjector. Participants were administered a single SC dose in upper arm, abdomen or thigh.
- Liquid Safety Syringe: Participants were administered 100 mg/mL SC dose of mepolizumab liquid formulation via disposable pre-filled safety syringe. Participants were administered a single SC dose in upper arm, abdomen or thigh.
Period: Overall Study
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Started | 85 | 79 | 80
Completed | 84 | 79 | 80
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Subjects (Safety) comprised of all participants who received mepolizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe | Total
Number analyzed (Participants) | 85 | 79 | 80 | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (15.06) | 46.5 (15.00) | 47.5 (14.94) | 46.7 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 38 | 114
  Male | 45 | 43 | 42 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 18 | 15 | 18 | 51
  American Indian or Alaska native | 1 | 0 | 0 | 1
  Central/South Asian heritage | 1 | 0 | 0 | 1
  East Asian heritage | 0 | 1 | 0 | 1
  Native Hawaiian or other pacific islander | 0 | 1 | 0 | 1
  Arabic/ North African heritage | 0 | 0 | 1 | 1
  White/Caucasian/European heritage | 64 | 61 | 61 | 186
  Asian and White | 0 | 1 | 0 | 1
  Black or African American and White | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Mepolizumab
Description: Blood samples were collected at indicated time points. Cmax following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with reconstituted lyophilized drug product from the vial. Pharmacokinetic (PK) Population comprised of all participants receiving study drug for whom a pharmacokinetic sample was obtained and analyzed.
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
micrograms per milliliter (µg/mL) | 11.57 (27.43) | 11.98 (24.96) | 12.07 (27.29)
Statistical Analysis 1: Comparison: Lyophilized Vial vs Liquid Autoinjector; Test type: Equivalence — Interpretation of the comparability of the autoinjector and safety syringe with the reconstituted lyophilized drug product was guided by a two-sided 90% confidence interval (CI) for the ratio of the geometric mean of test treatment to reference treatment in the range (0.80, 1.25) for Cmax; Ratio = 1.04, 90% CI 2-sided [0.98 to 1.11] — Ratio (autoinjector/lyophilized drug) for Cmax has been presented
Statistical Analysis 2: Comparison: Lyophilized Vial vs Liquid Safety Syringe; Test type: Equivalence — Interpretation of the comparability of the autoinjector and safety syringe with the reconstituted lyophilized drug product was guided by a two-sided 90% CI for the ratio of the geometric mean of test treatment to reference treatment in the range (0.80, 1.25) for Cmax; Ratio = 1.06, 90% CI 2-sided [0.99 to 1.12] — Ratio (safety syringe/lyophilized drug) for Cmax has been presented

2. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-t]), AUC From Time Zero Extrapolated to Infinite Time (AUC[0-inf]) of Mepolizumab
Description: Blood samples were collected at indicated time points. AUC(0-t) and AUC(0-inf) following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with lyophilized drug product. Fixed effects analysis of covariance model was used for analysis. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*µg/mL
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
Days*µg/mL
  AUC(0-t), n=85, 79, 80 | 403.84 (25.84) | 434.49 (22.62) | 415.15 (27.25)
  AUC(0-inf), n=84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  AUC(0-inf), n=84, 79, 80 | 450.83 (25.65) | 478.06 (24.76) | 454.11 (28.88)
Statistical Analysis 1: Comparison: Lyophilized Vial vs Liquid Autoinjector; Test type: Equivalence — Interpretation of the comparability of the autoinjector and safety syringe with the reconstituted lyophilized drug product was guided by a two-sided 90% CI for the ratio of the geometric mean of test treatment to reference treatment in the range (0.80, 1.25) for AUC (0-t); Ratio = 1.08, 90% CI 2-sided [1.01 to 1.15] — Ratio (autoinjector/lyophilized drug) for AUC(0-t) has been presented
Statistical Analysis 2: Comparison: Lyophilized Vial vs Liquid Safety Syringe; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 1.04, 90% CI 2-sided [0.97 to 1.12] — Ratio (safety syringe/lyophilized drug) for AUC(0-t) has been presented
Statistical Analysis 3: Comparison: Lyophilized Vial vs Liquid Autoinjector; Test type: Equivalence — Interpretation of the comparability of the autoinjector and safety syringe with the reconstituted lyophilized drug product was guided by a two-sided 90% CI for the ratio of the geometric mean of test treatment to reference treatment in the range (0.80, 1.25) for AUC (0-inf); Ratio = 1.07, 90% CI 2-sided [1.00 to 1.13] — Ratio (autoinjector/lyophilized drug) for AUC(0-inf) has been presented
Statistical Analysis 4: Comparison: Lyophilized Vial vs Liquid Safety Syringe; Test type: Equivalence — [test comment as in outcome 2, analysis 3]; Ratio = 1.02, 90% CI 2-sided [0.95 to 1.09] — Ratio (safety syringe/lyophilized drug) for AUC(0-inf) has been presented

3. Secondary Outcome: Time to Cmax (Tmax) and Last Time Point Where the Concentration is Above the Limit of Quantification (Tlast) of Mepolizumab
Description: Blood samples were collected at indicated time points. Tmax and tlast following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with lyophilized drug product.
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Median (Full Range); unit: Days
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
Days
  tmax | 7.04 [0.9 to 14.1] | 7.05 [2.9 to 21.0] | 7.06 [1.9 to 14.0]
  tlast | 83.97 [14.0 to 87.0] | 83.98 [81.1 to 87.1] | 83.99 [55.9 to 87.9]

4. Secondary Outcome: Apparent Clearance (CL/F) of Mepolizumab
Description: Blood samples were collected at indicated time points . CL/F following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with lyophilized drug product. Only those participants with data available were analyzed.
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/h)
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Liters per hour (L/h) | 0.009242 (27.91) | 0.008716 (28.74) | 0.009175 (39.30)

5. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Mepolizumab
Description: Blood samples were collected at indicated time points. Vd/F following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with lyophilized drug product. Only those participants with data available were analyzed.
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Liters (L) | 7.02 (22.49) | 6.74 (26.34) | 6.94 (31.84)

6. Secondary Outcome: Terminal Phase Elimination Rate Constant (Lambda z) of Mepolizumab
Description: Blood samples were collected at indicated time points. Lambda z following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with lyophilized drug product. Only those participants with data available were analyzed.
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hours
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Per hours | 0.0013157 (21.51) | 0.0012930 (26.20) | 0.0013228 (26.71)

7. Secondary Outcome: Terminal Phase Half-life (t½) of Mepolizumab
Description: Blood samples were collected at indicated time points for calculating t½. t½ following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with lyophilized drug product. Only those participants with data available were analyzed.
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Days | 21.95 (18.66) | 22.34 (21.38) | 21.83 (21.62)

8. Secondary Outcome: Percentage of AUC(0-inf) Obtained by Extrapolation (% AUCex) of Mepolizumab
Description: Blood samples were collected at indicated time points. Percentage AUCex following a single dose administration of liquid mepolizumab using a safety syringe and an autoinjector were compared with lyophilized drug product. Only those participants with data available were analyzed.
Time Frame: Day 1 (pre-dose, 2 hours, and 8 hours post-dose), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57 and 85 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Percentage | 7.67 (42.06) | 7.64 (47.30) | 7.20 (48.24)

9. Secondary Outcome: Number of Participants With On-treatment Non-serious Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or events associated with liver injury and impaired liver function were categorized as SAE. All Treated Subjects (Safety) comprised of all participants who received mepolizumab. Participants with non-serious AEs (3 percentage threshold) and SAEs has been reported.
Time Frame: Up to 28 days post-dose
Population: All Treated Subjects (Safety) Population
Measure: Number; unit: Participants
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
Participants
  Non-serious AEs | 11 | 13 | 14
  SAEs | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With On-treatment Systemic Reactions and Injection Site Reactions
Description: Adverse events of special interest like local injection site reactions and systemic reactions like allergic Type I hypersensitivity were reported along with AEs and SAEs. Participants with local injection site reaction and Allergic Type I hypersensitivity systemic reactions are reported here.
Time Frame: Up to 28 days post-dose
Population: All Treated Subjects (Safety) Population
Measure: Number; unit: Participants
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
Participants
  Systemic reactions | 0 | 0 | 0
  Injection site reactions | 1 | 1 | 2

11. Secondary Outcome: Number of Participants With Hematology Parameters Shifts From Baseline Relative to Normal Range
Description: Hematology parameters included assessment of platelet count, erythrocytes, leukocytes, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), neutrophils, lymphocytes, monocytes, eosinophils, basophils, hemoglobin and hematocrit. Participants were counted in the worst case category that their value changes to Low, Normal or High. Participants whose value category was unchanged or whose value became normal, were recorded in the "To Normal or No Change" category. The worst case post-Baseline values has been reported. For basophils the "to low" category is not applicable (NA) as the lower limit of normal is zero for this parameter.
Time Frame: Up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Number; unit: Participants
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
Participants
  Basophils, To low | NA — For basophils the "to low" category is not applicable (NA) as the lower limit of normal is zero for this parameter. | NA — For basophils the "to low" category is not applicable (NA) as the lower limit of normal is zero for this parameter. | NA — For basophils the "to low" category is not applicable (NA) as the lower limit of normal is zero for this parameter.
  Basophils, To normal or no change | 85 | 79 | 80
  Basophils, To high | 0 | 0 | 0
  Eosinophils, To low | 58 | 46 | 55
  Eosinophils, To normal or no change | 27 | 33 | 24
  Eosinophils, To high | 0 | 0 | 1
  Hematocrit, To low | 8 | 6 | 4
  Hematocrit, To normal or no change | 76 | 72 | 75
  Hematocrit, To high | 1 | 1 | 1
  Hemoglobin, To low | 12 | 8 | 13
  Hemoglobin, To normal or no change | 73 | 70 | 67
  Hemoglobin, To high | 0 | 1 | 0
  Lymphocytes, To low | 2 | 0 | 1
  Lymphocytes, To normal or no change | 83 | 79 | 79
  Lymphocytes, To high | 0 | 0 | 0
  MCH, To low | 0 | 5 | 2
  MCH, To normal or no change | 84 | 74 | 78
  MCH, To high | 1 | 0 | 0
  MCV, To low | 1 | 0 | 1
  MCV, To normal or no change | 83 | 79 | 79
  MCV, To high | 1 | 0 | 0
  Monocytes, To low | 11 | 8 | 12
  Monocytes, To normal or no change | 74 | 71 | 68
  Monocytes, To high | 0 | 0 | 0
  Neutrophils, To low | 7 | 11 | 9
  Neutrophils, To normal or no change | 77 | 68 | 71
  Neutrophils, To high | 1 | 0 | 0
  Platelets, To low | 0 | 0 | 1
  Platelets, To normal or no change | 85 | 78 | 79
  Platelets, To high | 0 | 1 | 0
  Erythrocytes, To low | 4 | 0 | 3
  Erythrocytes, To normal or no change | 81 | 78 | 77
  Erythrocytes, To high | 0 | 1 | 0
  Leukocytes, To low | 11 | 9 | 8
  Leukocytes, To normal or no change | 73 | 70 | 72
  Leukocytes, To high | 1 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters Shifts From Baseline Relative to Normal Range
Description: Blood samples were collected to evaluate clinical chemistry parameters, which included assessment of creatinine, creatine kinase, glucose, protein, potassium, urea, sodium, calcium, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), direct bilirubin (D.bili) and bilirubin, and albumin. Participants were counted in the worst case category that their value changes to Low, Normal or High. Participants whose value category was unchanged or whose value became normal, were recorded in the "To Normal or No Change" category. The worst case post-Baseline values has been reported. Only those participants with data available at the specified data points were analyzed. For the category "to low " NA indicates data was not available as the lower limit of normal is zero for this parameter.
Time Frame: Up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Number; unit: Participants
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Participants
  Glucose, To low | 1 | 0 | 0
  Glucose, To normal or no change | 83 | 79 | 80
  Glucose, To high | 0 | 0 | 0
  Albumin, To low | 0 | 0 | 0
  Albumin, To normal or no change | 83 | 79 | 80
  Albumin, To high | 1 | 0 | 0
  ALP, To low | 0 | 0 | 0
  ALP, To normal or no change | 84 | 79 | 80
  ALP, To high | 0 | 0 | 0
  ALT, To low | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter
  ALT, To normal or no change | 84 | 78 | 80
  ALT, To high | 0 | 1 | 0
  AST, To low | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter
  AST, To normal or no change | 84 | 78 | 80
  AST, To high | 0 | 1 | 0
  D.bilirubin, To low | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter
  D.bilirubin, To normal or no change | 83 | 79 | 80
  D.bilirubin, To high | 1 | 0 | 0
  Bilirubin, To low | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter
  Bilirubin, To normal or no change | 82 | 79 | 78
  Bilirubin, To high | 2 | 0 | 2
  Calcium, To low | 0 | 0 | 0
  Calcium, To normal or no change | 83 | 79 | 79
  Calcium, To high | 1 | 0 | 1
  Creatine kinase, To low | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter | NA — NA indicates data was not available as the lower limit of normal is zero for this parameter
  Creatine kinase,To normal or no change | 76 | 68 | 70
  Creatine kinase, To high | 8 | 11 | 10
  Creatinine, To low | 4 | 4 | 1
  Creatinine, To normal or no change | 79 | 75 | 79
  Creatinine, To high | 1 | 0 | 0
  Potassium, To low | 0 | 0 | 0
  Potassium, To normal or no change | 84 | 79 | 80
  Potassium, To high | 0 | 0 | 0
  Protein, To low | 1 | 1 | 0
  Protein, To normal or no change | 83 | 78 | 80
  Protein, To high | 0 | 0 | 0
  Sodium, To low | 1 | 0 | 0
  Sodium, To normal or no change | 83 | 79 | 80
  Sodium, To high | 0 | 0 | 0
  Urea, To low | 1 | 2 | 1
  Urea, To normal or no change | 83 | 75 | 79
  Urea, To high | 0 | 2 | 0

13. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured in supine position after 5 minutes rest. Baseline values for each assessment was the latest available assessment prior to receiving the single dose of mepolizumab. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
Millimeter of mercury (mmHg)
  DBP, Day 2, n=85, 79, 80 | 1.9 (7.36) | 3.1 (6.90) | 3.0 (6.47)
  DBP, Day 3, n=85, 79, 79: number analyzed (Participants) | 85 | 79 | 79
  DBP, Day 3, n=85, 79, 79 | 0.2 (7.06) | 1.7 (6.60) | 0.8 (7.90)
  DBP, Day 4, n=85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  DBP, Day 4, n=85, 78, 80 | 0.7 (6.44) | 1.6 (7.55) | 0.8 (6.33)
  DBP, Day 5, n=85, 79, 80 | 1.2 (7.04) | 2.4 (7.48) | 1.8 (6.40)
  DBP, Day 6, n=85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  DBP, Day 6, n=85, 78, 80 | 0.8 (6.80) | 0.9 (7.11) | 0.2 (7.96)
  DBP, Day 7, n=85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  DBP, Day 7, n=85, 78, 80 | 0.4 (7.44) | 0.3 (6.70) | 1.2 (7.50)
  DBP, Day 43, n=84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  DBP, Day 43, n=84, 79, 80 | 0.9 (8.04) | 2.2 (6.70) | 1.3 (7.22)
  DBP, Follow up, n=84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  DBP, Follow up, n=84, 79, 80 | 3.3 (8.26) | 3.5 (6.69) | 2.3 (6.70)
  SBP, Day 2, n=85, 79, 80 | 3.1 (10.61) | 2.0 (11.15) | 3.5 (11.25)
  SBP, Day 3, n=85, 79, 79: number analyzed (Participants) | 85 | 79 | 79
  SBP, Day 3, n=85, 79, 79 | 2.4 (10.45) | 0.7 (10.28) | 1.3 (11.12)
  SBP, Day 4, n=85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  SBP, Day 4, n=85, 78, 80 | 1.7 (9.51) | 1.7 (9.95) | 0.7 (10.07)
  SBP, Day 5, n=85, 79, 80 | 2.1 (11.03) | 2.5 (10.39) | 1.3 (9.67)
  SBP, Day 6, n=85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  SBP, Day 6, n=85, 78, 80 | 1.1 (9.38) | -0.6 (9.72) | -0.2 (10.81)
  SBP, Day 7, n=85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  SBP, Day 7, n=85, 78, 80 | 1.1 (10.95) | 0.1 (10.37) | 1.4 (11.30)
  SBP, Day 43, n=84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  SBP, Day 43, n=84, 79, 80 | 2.5 (11.21) | 2.2 (10.70) | 0.3 (11.93)
  SBP, Follow up, n=84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  SBP, Follow up, n=84, 79, 80 | 5.7 (10.21) | 3.8 (11.93) | 2.9 (11.67)

14. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in supine position after 5 minutes rest. Baseline values for each assessment was the latest available assessment prior to receiving the single dose of mepolizumab. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
Beats per minute
  Day 2, n=85, 79, 80 | 5.3 (9.19) | 5.6 (7.03) | 6.1 (9.78)
  Day 3, n= 85, 79, 79: number analyzed (Participants) | 85 | 79 | 79
  Day 3, n= 85, 79, 79 | 4.5 (8.01) | 5.0 (8.85) | 5.0 (9.37)
  Day 4, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 4, n= 85, 78, 80 | 3.7 (8.57) | 3.9 (7.93) | 3.2 (8.06)
  Day 5, n= 85, 79, 80 | 1.0 (9.02) | 1.0 (7.58) | 1.0 (8.73)
  Day 6, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 6, n= 85, 78, 80 | 2.4 (8.81) | 3.4 (8.46) | 4.3 (9.53)
  Day 7, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 7, n= 85, 78, 80 | 3.6 (9.05) | 2.5 (8.15) | 3.6 (10.33)
  Day 43, n= 84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  Day 43, n= 84, 79, 80 | 3.6 (10.29) | 3.7 (7.83) | 3.7 (10.77)
  Follow up, n= 84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  Follow up, n= 84, 79, 80 | 0.8 (10.56) | 1.0 (8.47) | 0.8 (8.91)

15. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured in supine position after 5 minutes rest. Baseline values for each assessment was the latest available assessment prior to receiving the single dose of mepolizumab. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
degree Celsius
  Day 2, n=85, 79, 80 | 0.08 (0.362) | 0.08 (0.389) | 0.01 (0.273)
  Day 3, n=85, 79, 79: number analyzed (Participants) | 85 | 79 | 79
  Day 3, n=85, 79, 79 | 0.09 (0.392) | 0.07 (0.310) | -0.02 (0.272)
  Day 4, n=85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 4, n=85, 78, 80 | 0.04 (0.289) | 0.05 (0.329) | -0.01 (0.293)
  Day 5, n=85, 79, 80 | -0.02 (0.264) | -0.02 (0.335) | -0.04 (0.317)
  Day 6, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 6, n= 85, 78, 80 | 0.01 (0.347) | 0.05 (0.350) | 0.00 (0.332)
  Day 7, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 7, n= 85, 78, 80 | 0.02 (0.281) | 0.10 (0.348) | 0.07 (0.280)
  Day 43, n= 84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  Day 43, n= 84, 79, 80 | 0.04 (0.300) | 0.06 (0.340) | -0.01 (0.293)
  Follow up, n= 84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  Follow up, n= 84, 79, 80 | 0.02 (0.296) | 0.02 (0.364) | 0.02 (0.280)

16. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in supine position after 5 minutes rest. Baseline values for each assessment was the latest available assessment prior to receiving the single dose of mepolizumab. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 85 | 79 | 80
breaths per minute
  Day 2, n= 85, 79, 80 | 0.0 (1.90) | 0.3 (2.30) | 0.5 (2.15)
  Day 3, n= 85, 79, 79: number analyzed (Participants) | 85 | 79 | 79
  Day 3, n= 85, 79, 79 | -0.2 (2.44) | 0.3 (2.60) | 0.1 (2.36)
  Day 4, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 4, n= 85, 78, 80 | -0.5 (2.09) | 0.4 (2.35) | 0.1 (2.10)
  Day 5, n= 85, 79, 80 | -0.2 (2.16) | 0.0 (2.80) | 0.2 (2.42)
  Day 6, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 6, n= 85, 78, 80 | -0.1 (2.03) | 0.2 (2.20) | 0.5 (2.45)
  Day 7, n= 85, 78, 80: number analyzed (Participants) | 85 | 78 | 80
  Day 7, n= 85, 78, 80 | -0.2 (2.02) | 0.1 (2.23) | 0.2 (2.06)
  Day 43, n= 84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  Day 43, n= 84, 79, 80 | 0.3 (2.03) | 0.4 (2.14) | 0.3 (2.07)
  Follow up, n= 84, 79, 80: number analyzed (Participants) | 84 | 79 | 80
  Follow up, n= 84, 79, 80 | -0.1 (2.17) | 0.6 (2.11) | 0.5 (2.07)

17. Secondary Outcome: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings
Description: Single measurements of 12-lead ECGs were obtained after 5 minutes of rest in a supine position for the participant. ECG was performed on Day 1 and Day 85 using an automated ECG machine. Baseline values for each assessment was the latest available assessment prior to receiving the single dose of mepolizumab. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Participants with abnormal ECG findings that are clinically not significant and clinically significant data has been presented here. The data of worst case post-Baseline is presented here. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline and Day 85
Population: All Treated Subjects (Safety) Population
Measure: Number; unit: Participants
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Participants
  Abnormal not clinically significant | 15 | 16 | 19
  Abnormal clinically significant | 1 | 0 | 1

18. Secondary Outcome: Number of Participants With Positive Anti-mepolizumab Binding Antibodies
Description: Blood samples were collected for the determination of anti-mepolizumab antibodies. A binding anti-drug antibody (ADA) assay was performed. There were three tiered analysis: screening, confirmation and titration. The results of binding ADA were categorized as negative, transient positive (defined as a single confirmatory positive immunogenic response that does not occur at the final study assessment) or persistent positive (defined as a confirmatory positive immunogenic response for at least 2 consecutive assessments excluding the Screening visit, or a single result at the final study assessment). A participant was considered positive if they had at least one positive post-Baseline ADA result. Number of participants with positive anti-mepolizumab antibodies at any time post-Baseline are presented here. Only those participants available at the specified time points were analyzed.
Time Frame: Up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Number; unit: Participants
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 84 | 79 | 80
Participants
  Transient positive | 1 | 1 | 0
  Persistent positive | 2 | 4 | 3

19. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies
Description: Blood samples were collected for the determination of positive neutralizing antibodies. A neutralizing antibody assay was performed. Neutralizing antibody test was only carried out for participants who have had a positive confirmatory binding antibody test result at visit. A participant was considered positive if they had at least one positive post-Baseline neutralizing antibody result. Number of participants with positive neutralizing antibodies at any time post-Baseline are presented here. Only those participants available at the specified time points were analyzed.
Time Frame: Up to Day 85
Population: All Treated Subjects (Safety) Population
Measure: Number; unit: Participants
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
Number analyzed (Participants) | 3 | 5 | 3
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and up to 28 days post-dose.
Description: All Treated Subjects (Safety) comprised of all participants who received mepolizumab.
Arm/Group | Lyophilized Vial | Liquid Autoinjector | Liquid Safety Syringe
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/79 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/79 | 0/80
Other Adverse Events (participants affected / at risk) | 11/85 | 13/79 | 14/80
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyophilized Vial (N=85) | Liquid Autoinjector (N=79) | Liquid Safety Syringe (N=80)
Headache (Nervous system disorders) | 6 (6) | 9 (9) | 8 (9)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 6 (6)
Fatigue (General disorders) | 5 (5) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03014674/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03014674/SAP_001.pdf